CLINICAL TRIAL: NCT00444119
Title: Survey in Patients With Chronic Adrenal Insufficiency in Germany
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Other Study IDs: Wü_NNRIS_45/04
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-03-07 (Estimated); Status verified 2007-03

CONDITIONS: Adrenal Insufficiency; Addison's Disease
Keywords: adrenal insufficiency; subjective health status; quality of life; adrenal crisis; hormone replacement; DHEA
MeSH Terms: conditions — Adrenal Insufficiency; Addison Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this survey is to assess patients with chronic primary or secondary adrenal failure regarding subjective health status, incidence and causes of adrenal crisis, hormone replacement regimens and concomitant endocrine or non endocrine disease.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* chronic adrenal failure with disease duration > 12 months and hormone replacement therapy for cortisol deficiency

Exclusion Criteria:

* adrenal insufficiency due to adrenocortical carcinoma
* AI due to long-term pharmacological glucocorticoid treatment
* glucocortiocid doses above 7.5 mg prednisolone equivalent for other reasons than AI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Principal Investigator — University of Wuerzburg
Locations (2):
- Germany (2):
  - Dept of Medicine, Gastroenterology, Hepatology and Endocrinology, Charité Campus Mitte, Charité, University Medicine Berlin, Berlin
  - University of Wuerzburg, Dept of Medicine - Endocrine and Diabetes unit, Würzburg

REFERENCES:
- [Derived] Hahner S, Loeffler M, Fassnacht M, Weismann D, Koschker AC, Quinkler M, Decker O, Arlt W, Allolio B. Impaired subjective health status in 256 patients with adrenal insufficiency on standard therapy based on cross-sectional analysis. J Clin Endocrinol Metab. 2007 Oct;92(10):3912-22. doi: 10.1210/jc.2007-0685. Epub 2007 Aug 7. PMID 17684047